CLINICAL TRIAL: NCT05830864
Title: Multicenter Retrospective Study of Isoflurane in Refractory and Super-Refractory Status Epilepticus (I-Seizure)
Brief Title: Multicenter Retrospective Study of Isoflurane in Refractory and Super-Refractory Status Epilepticus
Acronym: I-Seizure
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, Director of Clinical Research Unit, Hopital of Melun
Other Study IDs: MIR-2023-01
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Refractory Status Epilepticus
Keywords: Isoflurane
MeSH Terms: conditions — Status Epilepticus | interventions — Isoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main cohort: Adult patients with refractory status epilepticus treated by Isoflurane as third anticonvulsive therapy
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Isoflurane — no other intervention

SUMMARY:
Isoflurane might be used as anticonvulsive therapy in refractory status epilepticus. The aim of the study is to assess the efficiency of Isoflurane in this indication.

DETAILED DESCRIPTION:
Investigators will collect in 4 ICUs the data from consecutive patients hospitalized between january 2016 and january 2023. Included patient were those treated by Isoflurane for refractory status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, hospitalized in ICU between 2016-01-01 and 2023-01-01, suffering refractory status epilepticus treated by inhaled Isoflurane as third anticonvulsive therapy

Exclusion Criteria:

* post-anoxic refractory status epilepticus after cardiac arrest, withdrawal of consent for medical data use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with eligibility criteria in the sites of study will be included int the study
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
rate of crisis control | 3 months
  rate of patients with crisis control or complete awakening

CONTACTS AND LOCATIONS:
Overall Officials: SEBASTIEN JOCHMANS, MD, Study Director — GHSIF MELUN
Locations (4):
- France (4):
  - Ch Bethune Beuvry, Beuvry
  - CHU Brest, Brest
  - GH Sud Ile de France, Hôpital de Melun-Sénart, Melun
  - CH Toulon - Sainte Musse, Toulon

IPD SHARING:
Plan to Share IPD: Undecided
After study completion, on justified demand and after review board authorization

REFERENCES:
- [Background] Meiser A, Volk T, Wallenborn J, Guenther U, Becher T, Bracht H, Schwarzkopf K, Knafelj R, Faltlhauser A, Thal SC, Soukup J, Kellner P, Druner M, Vogelsang H, Bellgardt M, Sackey P; Sedaconda study group. Inhaled isoflurane via the anaesthetic conserving device versus propofol for sedation of invasively ventilated patients in intensive care units in Germany and Slovenia: an open-label, phase 3, randomised controlled, non-inferiority trial. Lancet Respir Med. 2021 Nov;9(11):1231-1240. doi: 10.1016/S2213-2600(21)00323-4. Epub 2021 Aug 26. PMID 34454654
- [Background] Stetefeld HR, Schaal A, Scheibe F, Nichtweiss J, Lehmann F, Muller M, Gerner ST, Huttner HB, Luger S, Fuhrer H, Bosel J, Schonenberger S, Dimitriadis K, Neumann B, Fuchs K, Fink GR, Malter MP; IGNITE Study Group, with support from the German Neurocritical Care Society (DGNI). Isoflurane in (Super-) Refractory Status Epilepticus: A Multicenter Evaluation. Neurocrit Care. 2021 Dec;35(3):631-639. doi: 10.1007/s12028-021-01250-z. Epub 2021 Jul 20. PMID 34286464